CLINICAL TRIAL: NCT00496340
Title: Phase II Trial of Pentostatin and Targeted Busulfan as a Novel Reduced Intensity Regimen for Allogeneic Hematopoietic Stem Cell Transplantation Using Laboratory-Guided (CD4-guided) Immunosuppression.
Brief Title: Phase II Trial of Pentostatin and Targeted Busulfan
Acronym: Pento & tBU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15009
Record Dates: First submitted 2007-06-29; First posted 2007-07-04 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-03

CONDITIONS: Hematologic Malignancies
Keywords: Pentostatin; Busulfan; Rituxan; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Pentostatin; Busulfan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Conditioning Followed by HCT (Experimental): Pentostatin/Busulfan/Rituximab/Allogeneic Hematopoietic Cell Transplant (HCT).
  Pre-conditioning therapy:
  All participants will receive pentostatin 4 mg/m^2 on day -28. Patients may receive additional doses on days -21 & -14 depending on cell counts.
  Conditioning:
  1. Patients will receive anti-seizure prophylaxis with lorazepam 0.5 mg every 6 hours beginning day -6.
  2. Intravenous Busulfan (1st dose) at a dose of 200mg/m^2 on day -4.
  3. Patient will then receive pentostatin at a dose of 4 mg/m^2 by intravenous infusion over 1-2 hours on days -4, -3.
  4. Intravenous Busulfan (2nd dose) will be administered on day (-2) to target a total AUC of 16,000 +/- 1600.
  5. Hematopoietic progenitor cells to be infused at least 36 hours after last dose of Busulfan.
  6. Rituximab: Patients with CD20+ expressing malignancies will be treated with rituximab at a dose of 375 mg/m^2 according to prescribing and institutional guidelines.
  Interventions: Drug: Pentostatin; Drug: Busulfan; Drug: Rituximab; Procedure: Allogeneic Hematopoietic Cell Transplant

INTERVENTIONS:
Drug: Pentostatin — Pre-conditioning therapy:
  All participants will receive pentostatin 4 mg/m^2 on day -28. Patients may receive additional doses on days -21 & -14 depending on cell counts.
  Participant will receive pentostatin at a dose of 4 mg/m^2 by intravenous infusion over 1-2 hours on days -4, -3.
  Other Names: deoxycoformycin
Drug: Busulfan — Pre-conditioning therapy:
  Intravenous Busulfan (1st dose) at a dose of 200mg/m^2 on day -4.
  Intravenous Busulfan (2nd dose) will be administered on day (-2) to target a total AUC of 16,000 +/- 1600.
  Other Names: BU; Busulfex
Drug: Rituximab — Pre-conditioning therapy:
  Patients with CD20+ expressing malignancies will be treated with rituximab at a dose of 375 mg/m^2 according to prescribing and institutional guidelines.
  Other Names: Rituxan
Procedure: Allogeneic Hematopoietic Cell Transplant — Hematopoietic progenitor cells to be infused at least 36 hours after last dose of Busulfan.

SUMMARY:
The objective of this trial is to determine whether a regimen of pentostatin and busulfan (IV) can facilitate engraftment of human leukocyte antigen (HLA) partially compatible siblings and unrelated donor transplants by using CD4+ laboratory-guided immunosuppression among 41 transplant patients meeting the inclusion criteria.

DETAILED DESCRIPTION:
Pentostatin (deoxycoformycin) is a purine analogue that is currently indicated for the treatment of chemo-naïve or interferon-refractory hairy cell leukemia. Pentostatin represents an ideal agent for conditioning recipients before allogeneic hematopoietic cell transplantation (HCT) due to its significant effect on lymphocytes and relatively reduced myelosuppression as compared to other purine analogues. It is a potent inhibitor of the enzyme adenosine deaminase (ADA) whose activity is generally more pronounced in T lymphocytes as compared to their B counterparts. Also, pentostatin has been shown, though its immunomodulatory effect to be active in patients with steroid-refractory acute graft versus host disease (aGVHD).

Pentostatin-based regimens have been studied as a conditioning strategy for patients undergoing allogeneic stem cell transplantation. Chan et al. evaluated 18 myelodysplastic syndrome (MDS) patients ineligible for standard allogeneic transplantation. In that series, patients received conditioning with a preparative regimen of photopheresis day -7 and -6, pentostatin 4 mg/m^2 by continuous infusion day -5 and -4, and total body irradiation 600 centigray (cGy) in 3 fractions day -3 and -2, followed by allogeneic stem cell infusion from 6/6 or 5/6 HLA-matched related donors or 6/6 HLA-matched unrelated donors. Sixteen of 18 (89%) patients developed full donor chimerism, with no day +100 transplant-related mortality (TRM). Grade 2 to 4 aGVHD and extensive chronic graft versus host disease (GVHD) developed in 19% and 18% of patients, respectively. Disease relapse occurred in 2 patients. At a median follow-up of 14 months (range, 1-35 months), the 1-year failure-free and overall survival were 64% and 65%, respectively. These findings clearly suggest that Pentostatin-based regimens are capable of achieving a successful donor engraftment and durable disease-remission with significantly lesser transplant toxicity and grade 2 to 4 acute GVHD. Pavletic et al., demonstrated that Pentostatin induces significant lympho-depleting effects with a promising safety, supporting its use as a conditioning regimen in non-myeloablative strategies with hematopoietic cell infusions as early as 7 days after initiation of Pentostatin.

Busulfan was available primarily as an oral formulation until recently. The oral drug has variable bioavailability that has been linked to erratic gastrointestinal absorption from patient to patient. In a phase I trial, Andersson et al evaluated an IV Bu formulation using dimethylacetamide and PEG400 as the solvent. This is the formulation currently marketed in the USA (Busulfex ESP Pharma). Fifteen patients with advanced hematologic malignancies were treated with BU every 6 hours for a total of 16 doses followed by cyclophosphamide (CY) 60mg/kg for 2 doses and hematopoietic cell transplant. The first BU dose given was by IV. The starting IV dose was 0.08mg/kg which was then escalated to 0.2, 0.4, and finally to 0.8mg/kg in cohorts of 3 patients each. Six hours after the start of the IV BU infusion, the patients began to receive oral BU 1mg/kg every 6 hours for 15 doses. Pharmacokinetic profiles were obtained to determine an equivalent exposure of IV BU to the oral BU dose of 1mg/kg. It was noted that the toxicity profile and rates of engraftment were similar to that of the oral drug (i.e., no additional toxicities were found attributable to the solvents). An IV dose of 0.8mg/kg gave an equivalent AUC (but with less variability) as the oral dose of 1mg/kg with a mean AUC of 1189 micrometer (uM)-min (range 964-1547uM-min; 24h DIE 4756uM-min [range 3856-6188uM-min]). Thus, 0.8mg/kg was chosen by the investigators as the dose to proceed to phase II testing. A subsequent phase II multicenter trial in 61 patients with a variety of hematologic malignancies using 0.8mg/kg every 6 hours x 16 doses of IV BU and 120mg/kg CY prior to hematopoietic stem cell transplant. Pharmacokinetic analyses were also done. Once again, it was shown that the toxicity and outcome data was similar to that published for the oral BU. There were no patients with seizures. Lung toxicities occurred in two patients, one with diffuse alveolar hemorrhage (DAH) and one with interstitial pneumonitis (IP); the latter patient had a history of lung irradiation. Grade 1-2 nausea and emesis occurred in 43% and grade 3 in 7%. Mucositis was grade 2 in 44%, Grade 3 in 26% and lasted a median of 6 days. There were five (8%) cases of veno-occlusive disease (VOD), which was fatal in two (3%). Treatment related mortality at 100 days was 9.8%. The AUC was <1500 uM-min (24h DIE <6000uM-min) in 55%; 86% of patients maintained an AUC between 800 and 1500uM-min (24h DIE 3200-6000uM-min). The AUC at dose 1 and dose 9 were similar indicating a consistent dose-to-dose behavior. The authors concluded that IV BU in this setting was well tolerated and demonstrated excellent antitumor efficacy, likely resulting from predictable pharmacokinetics. Based on these and other studies, IV administration has become the preferred route for BU when given in the high dose transplant setting. Fernandez, et al. evaluated the use of IV Bu (Busulfex® ESP Pharma) in either a once daily or twice daily dosing schedule when given as a part of BUCY regimen (BU: 3.2 mg/kg and CY 120mg/kg) prior to transplant. In both dosing schedules, there was little variability in the dose-to-dose levels and the pharmacokinetics of the first dose could predict the data on subsequent doses. In the twice-daily group, AUC 3390uM-min (2400- 4678uM-min; 24h DIE 6780uM-min [4800-9356uM-min]) and the once daily group the AUC 5561uM-min (4412 - 7368uM-min). The pharmacokinetic profiles (AUC, CL, Cmax and t 1/2) were similar from dose to dose. In the twelve patients studied, the following grade 3 toxicities were reported: mucositis, anorexia, infection, epistaxis and hyperglycemia. Two patients died: one from sepsis from presumed fungal infection and one sudden cardiac death. One patient developed mild, reversible VOD. Daily dosing of IV Bu results in similar outcomes and toxicity profile compared to oral dosing and ease in delivering a targeted exposure of BU. The importance of being able to target BU exposure has been illustrated in the above discussion of reports correlating BU pharmacokinetic parameters with its toxicity and efficacy. Thus, by utilizing a once daily IV dose, targeted to prespecified levels, BU therapy can be optimized to limit toxicity and maximize efficacy.

To see if the AUC of IV Bu was correlated to adverse effects, Andersson and colleagues treated 36 chronic myelogenous leukemia (CML) patients with either fixed or adjusted dose BuCy. The first 25 patients were given a fixed dose of Bu 0.8mg/kg every 6 hours. In the subsequent 12 patients, doses were adjusted to achieve an AUC of 1250uM-min (24h DIE 5000uM-min). At steady state, the population median AUC was 1265uM-min (range, 816-1905uM-min [24h DIE 5056uM-min; 3264-7620uM-min]). They found that the probabilities of developing gastrointestinal toxicity, hepatotoxicity, mucositis, and acute GVHD all increased with increasing AUC. The 26 patients within AUC of 950 - 1520uM-min (24h DIE 3800-6080uM-min) had a decreased incidence of death compared with the 10 patients outside this range. There were no cases of hepatic veno-occlusive disease or seizures. These were small numbers but did indicate a trend towards achieving an optimal systemic exposure by delivering individualized doses and a suggestion of a "therapeutic window" for Bu in this setting. The importance of being able to target BU exposure has been illustrated in the above discussion of reports correlating Bu pharmacokinetic parameters with its toxicity and efficacy. Thus, by utilizing a once daily IV dose, targeted to prespecified levels, Bu therapy can be optimized to limit toxicity and maximize efficacy.

Rituximab is an anti-CD20 human-mouse chimeric monoclonal antibody indicated for the treatment of relapsed or refractory, low-grade or follicular, CD20-positive, B-cell NHL. The use of rituximab, as monotherapy, results in significant responses and durations of response in patients with indolent non-Hodgkin's lymphoma (NHL); its efficacy improves even further when used in combination with chemotherapy for both indolent and aggressive NHL. Responses to rituximab treatment vary by the histologic subtype of NHL. In patients with low-grade follicular lymphoma, response rates are approximately 70% to 75% with first-line therapy. On the other hand, patients with diffuse B-cell large-cell lymphoma (DBLCL), single-agent rituximab results in response rates of 30% to 40% have been reported. Rituximab significantly increases response rates when used in combination with cyclophosphamide, doxorubicin, vincristine, and prednisone.

CD20 is not expressed by hematopoietic stem cells, and therefore, we hypothesize that treatment with rituximab is safe and would not inhibit engraftment produced by these early progenitors. Treatment with rituximab may successfully eliminate minimal residual disease, further delaying or preventing disease relapse and potentially extending the duration of survival in CD20+ expressing malignancies.

ELIGIBILITY:
Inclusion Criteria:

Recipients:

* Age: greater than 18 years of age, or younger with parental consent.
* HLA A, B, C, DRB1, DQB1, 10/10 or 9/10 allele sequence matched related donor or unrelated donor available
* Histologically confirmed diagnosis by pathologic review.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1, or Karnofsky performance status of greater than 70
* Organ function:

  1. Pulmonary: diffusing capacity of lung for carbon monoxide (DLCO) >/= 50%
  2. Cardiac: left ventricular ejection fraction >/= 50%
  3. Renal: creatinine clearance (measured or calculated) equal or greater than 50 ml/min (at any time pentostatin is administered)
  4. Hepatic: total bilirubin less than or equal to 2mg/dL, (Gilbert and other syndromes with increased indirect bilirubin should be allowed); serum transaminases less than two times the institutional upper limit of normal (< 2 x ULN).

Donors:

* Capable of receiving Granulocyte Colony-Stimulating Factor (G-CSF) and undergo apheresis
* Age >18
* Signed informed consent form in accordance with institutional or National Donor Marrow Program (NMDP) policies

Exclusion Criteria:

Recipients:

* Pregnant or lactating women
* HIV or seropositive, confirmed by nucleic acid test (NAT)
* Active central nervous system (CNS) malignancy
* Active infection
* Unfavorable psychosocial evaluation or history of poor compliance to prescribed medical care.
* Current use of metronidazole or acetaminophen; patients must discontinue use of these agents at least 7 days prior to the start of Busulfex administration
* Prior allogeneic HCT (patients who had received a prior autologous HCT will be allowed)
* Lack of a capable caregiver.
* Presence of any of the following comorbid conditions

  1. History of recent myocardial infarction within 30 days
  2. Congestive heart failure (NY class III, IV or if symptomatically uncontrolled)
  3. Peripheral vascular disease (including intermittent claudication or history of bypass for arterial insufficiency)
  4. Untreated thoracic or abdominal aneurysm (6 cm or more)
  5. History of any cerebrovascular accident including transient ischemic attacks within 30 days
  6. Dementia
  7. History of recent gastrointestinal bleeding (within 30 days)
  8. Connective tissue/rheumatologic disorders
  9. Hemiplegia/paraplegia
  10. History of solid tumor excluding skin or cervical carcinoma after curative resection. Patients with other prior solid tumor (s) who are in remission for more than 5 years will be allowed on a case-by-case basis

Donors:

* Pregnant or lactating women
* HIV seropositive, confirmed by NAT
* Human T- lymphotropic virus (HTLV) I/II seropositive
* Hepatitis B or C seropositive
* Donors with uncontrolled bacterial, viral, fungal or parasitic infections.
* Donors with known hypersensitivity to recombinant human G-CSF or any E. coli-derived products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-07; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcie Riches, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at H. Lee Moffitt Cancer Center between February 2008 and March 2011.
Groups:
- Conditioning Followed by HCT: Pentostatin/Busulfan/Rituximab/Allogeneic Hematopoietic Cell Transplant (HCT)
  Pre-conditioning therapy:
  All participants receive pentostatin 4 mg/m^2 on day -28, may receive additional doses on days -21 & -14 depending on cell counts.
  Conditioning:
  1. Anti-seizure prophylaxis with lorazepam 0.5 mg every 6 hours beginning day -6
  2. Intravenous Busulfan (1st dose) at a dose of 200mg/m^2 on day -4
  3. Pentostatin, 4 mg/m^2 by intravenous infusion over 1-2 hours on days -4, -3
  4. Intravenous Busulfan (2nd dose) on day (-2) to target a total area under curve (AUC) of 16,000 +/- 1600
  5. Hematopoietic progenitor cells infused at least 36 hours after last dose of Busulfan
  6. Patients with CD20+ expressing malignancies treated with rituximab at a dose of 375 mg/m^2 according to prescribing and institutional guidelines
Period: Overall Study
Arm/Group | Conditioning Followed by HCT
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants. Bone marrow chimerism data were available for only 38 patients at day +28 and for only 36 patients at day +100.
Groups:
- Conditioning Followed by HCT: Pentostatin/Busulfan/Rituximab/Allogeneic Hematopoietic Cell Transplant (HCT)
  Pre-conditioning therapy:
  All participants receive pentostatin 4 mg/m^2 on day -28, may receive additional doses on days -21 & -14 depending on cell counts.
  Conditioning:
  1. Anti-seizure prophylaxis with lorazepam 0.5 mg every 6 hours beginning day -6
  2. Intravenous Busulfan (1st dose) at a dose of 200mg/m^2 on day -4
  3. Pentostatin, 4 mg/m^2 by intravenous infusion over 1-2 hours on days -4, -3
  4. Intravenous Busulfan (2nd dose) on day (-2) to target a total AUC of 16,000 +/- 1600
  5. Hematopoietic progenitor cells infused at least 36 hours after last dose of Busulfan
  6. Patients with CD20+ expressing malignancies treated with rituximab at a dose of 375 mg/m^2 according to prescribing and institutional guidelines
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 53 [29 to 73]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Greater Than or Equal to 50% Donor Chimerism
Description: The primary endpoint was achievement of >/= 50% donor chimerism in CD3+ peripheral blood lymphocytes by day +28 (± 7) after allogeneic hematopoietic cell transplantation (allo-HCT).
Time Frame: 28 days post-transplant
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
percentage of participants | 100

2. Secondary Outcome: Cumulative Incidence of Hematopoietic Cell Engraftment
Description: Hematologic engraftment: defined as time to achieve an absolute neutrophil count (ANC) >/= 500/µl for 3 consecutive days or a platelet count of >/= 20,000//µl without the need for platelet support.
Time Frame: 28 days post-transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
percentage of participants | 97.6 [90.6 to 100]

3. Secondary Outcome: Rate of T-cell (CD3+) and Myeloid (CD33+) Chimerism by Day +28
Description: Median Percentage of Donor Cells in Study Population (Chimerism).
Time Frame: 28 days post-transplant
Population: Participants with bone marrow chimerism data available at time of analysis.
Measure: Median (95% Confidence Interval); unit: percentage of cells
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 38
percentage of cells
  CD3+ | 87 [61 to 100]
  CD33+ | 100 [95 to 100]

4. Secondary Outcome: Rate of T-cell (CD3+) and Myeloid (CD33+) Chimerism by Day +100
Description: Median Percentage of Donor Cells in Study Population (Chimerism).
Time Frame: 100 days post-transplant
Population: Participants with bone marrow chimerism data available at time of analysis.
Measure: Median (95% Confidence Interval); unit: percentage of cells
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 36
percentage of cells
  CD3+ | 96 [64 to 100]
  CD33+ | 100 [100 to 100]

5. Secondary Outcome: Non-relapse Mortality Rate (NRM)
Description: The cumulative incidence of NRM after allo-HCT.
Time Frame: Up to 2 years post-transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
percentage of participants
  Day +100 | 2 [0 to 9]
  2 Years | 17 [7 to 30]

6. Secondary Outcome: Incidence of Infections
Description: Infections: Incidence of infections (opportunistic and non-opportunistic) following conditioning.
Time Frame: Up to 2 years post-transplant
Population: All participants
Measure: Number; unit: participants
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
participants
  Cytomegalovirus (CMV) Reactivation | 17
  Epstein-Barr virus (EBV) Reactivation | 3
  Post-transplantation Lymphoproliferative Disorder | 1
  Viral Infections | 5
  Lung Infections | 2

7. Secondary Outcome: Time to Incidence of Graft Versus Host Disease (GVHD)
Description: The median time from allo-HCT to the initiation of tacrolimus (TAC) taper.
  The median time to onset of acute GVHD (aGVHD). Clinical manifestations of acute GVHD include a classic maculopapular rash; persistent nausea and/or emesis; abdominal cramps with diarrhea; and a rising serum bilirubin concentration.
Time Frame: Up to 2 years post-transplant
Population: All participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
days
  Initiation of TAC Taper | 62 [38 to 377]
  Onset of aGVHD | 33 [14 to 85]

8. Secondary Outcome: Incidence of Graft Versus Host Disease (GVHD)
Description: By day +100, the cumulative incidence of GVHD, acute of grades 2-4, and 3-4.
  At 2 years, the cumulative incidence of chronic GVHD of any severity according to National Institutes of Health (NIH) consensus criteria. Diagnosis of chronic GVHD requires the presence of at least one diagnostic clinical sign of chronic GVHD or the presence of at least one distinctive manifestation confirmed by pertinent biopsy or other relevant tests in the same or another organ. Furthermore, other possible diagnoses for clinical symptoms must be excluded. No time limit is set for the diagnosis of chronic GVHD.
  At 2 years, the cumulative incidence of moderate/severe chronic GVHD.
Time Frame: Up to 2 years post-transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
percentage of participants
  Day +100 aGVHD Grade 2-4 | 59 [43 to 75]
  Day +100 aGVHD Grade 3-4 | 19 [7 to 35]
  2 Years, Chronic GVHD of Any Severity | 69 [53 to 83]
  2 Years, Moderate/Severe Chronic GVHD | 58 [39 to 75]

9. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS)
Description: PFS at 2 years post-transplant. PFS, defined as time from day of hematopoietic cell infusion to disease relapse. Relapsed disease: Disease was in complete remission post-transplant but returned (e.g., >5% blast in bone marrow or any peripheral blasts).
Time Frame: 2 years post-transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
percentage of participants | 55 [39 to 69]

10. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: OS at 2 years post-transplant. OS, defined as time from day of hematopoietic cell infusion to death from any cause.
Time Frame: 2 years post-transplant
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Followed by HCT
Number analyzed (Participants) | 42
percentage of participants | 68 [53 to 81]

ADVERSE EVENTS:
Time Frame: Up to 2 years post-transplant
Description: There were no Adverse Events (AEs) that would not be expected for transplant patients.
Arm/Group | Conditioning Followed by HCT
Serious Adverse Events (participants affected / at risk) | 25/42
Other Adverse Events (participants affected / at risk) | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conditioning Followed by HCT (N=42)
Blood/Bone Marrow - Other, Complications with GVHD (Blood and lymphatic system disorders) | 1
Cardiac General - Other, Cardiac arrest (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Coagulation - Other, Right jugular vein occlusion (Blood and lymphatic system disorders) | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2
Fever (in the absence of neutropenia) (General disorders) | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 5
Dermatology/Skin - Other, Shingles reactivation (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Enteritis (inflammation of the small bowel) (Gastrointestinal disorders) | 1
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hematoma (Vascular disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 2
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Eye NOS (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Skin (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Upper airway (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Stomach (Infections and infestations) | 1
Creatinine - high (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1
Cervical spine-range of motion (Musculoskeletal and connective tissue disorders) | 1
Joint-effusion (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 2
Mental status (Psychiatric disorders) | 2
Seizure (Nervous system disorders) | 1
Vision-photophobia (Eye disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Pain - Other, chest/epigastric (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other, Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Obstruction, GU - Bladder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Secondary Malignancy - Basal cell (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Secondary Malignancy - EBV driven PTLD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Bone marrow chimerism data were available for only 38 patients at day +28 and for only 36 patients at day +100.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes